CLINICAL TRIAL: NCT03382197
Title: Regional Ventilation and Radioaerosol Pulmonary Deposition Through Different Positive Pressure Strategies in COPD Patients.
Brief Title: Different Positive Pressure Strategies in COPD Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Catarina Souza Ferreira Rattes Lima, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFPE_FISIO_RESP
Record Dates: First submitted 2017-12-06; First posted 2017-12-22 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: aerosol therapy; positive pressure; electrical impedance tomography; pulmonary scintigraphy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will be randomized regarding the order of intervention they will receive:
  Group 1 - control intervention, will only perform nebulization; Group 2 - intervention, will perform nebulization associated with positive expiratory pressure valve in the airways (EPAP); Group 3 - intervention, will perform nebulization associated with non-invasive ventilation Bi-level mode;
  All patients will be evaluated BEFORE, DURING and AFTER each intervention through Electrical Impedance Tomography, Pulmonary Scintigraphy and Spirometry.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Two experienced researchers will participate in the study, one being responsible for the evaluation of the outcomes (researcher 1) and the other responsible for the application of the intervention in each patient (researcher 2). The researcher 2 will receive in opaque and sealed envelopes the randomized order of the interventions of each patient, keeping them in secrecy until the end of the whole study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nebulization (Experimental): control intervention, will only perform nebulization;
  Interventions: Device: Nebulization
- Positive expiratory pressure valve (Experimental): Intervention, will perform nebulization associated with positive expiratory pressure valve in the airways (EPAP)
  Interventions: Device: Positive expiratory pressure valve
- Nonivasive ventilation (Experimental): intervention, will perform nebulization associated with non-invasive ventilation Bi-level mode;
  Interventions: Device: Nonivasive ventilation

INTERVENTIONS:
Device: Nebulization — For inhalation of the radioaerosol a dose of DTPA-Tc99m (methionine-labeled diethylnitriaminepentaacetic acid) with 1mCi activity, associated with 10 drops of Fenoterol Bromide and 20 drops of Ipatropium Bromide diluted for a total of up to 3 ml of saline solution 0.9%. A MESH vibrating nebulizer (NIVO, Philips Respironics, Murrysville, Pennsylvania) will be used.
  Arms: Nebulization
Device: Positive expiratory pressure valve — For nebulization associated with the EPAP valve will be used a non-invasive distribution system consisting of a non-toxic orofacial mask connected to a spring loaded EPAP valve. This mask will be secured to the patient's face through tabs in order to prevent leakage and to maintain proper pressurizing and better patient adaptation.
  Arms: Positive expiratory pressure valve
Device: Nonivasive ventilation — For nebulization associated with NIV, a noninvasive distribution system consisting of a non-toxic orofacial mask connected to the NIV circuit will be used, and the latter will be being fed by a radioaerosol flow generated by a nebulizer coupled to the circuit. This mask will be secured to the patient's face through tabs in order to prevent leakage and to maintain proper pressurizing and better patient adaptation.
  Arms: Nonivasive ventilation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by a poorly reversible airway obstruction and consequent systemic manifestations. Its high prevalence and high number of diagnosed patients has become a challenge for health services due to the costs of diagnosis and treatment of these patients. Positive pressure and aerosol therapy are preferred therapies for the management of COPD symptoms, but their effects when associated are poorly studied. The objective of this study is to compare the effects of different positive pressure strategies associated with aerosol therapy through Pulmonary Scintigraphy and Electrical Impedance Tomography (EIT) in patients with COPD in the intercrise period. This is a randomized, crossover, blinded and allocated crossover type clinical trial in which patients with moderate to severe COPD will be allocated to three intervention groups with different strategies for positive pressure associated with aerosol therapy: control group 1 nebulization), group 2 nebulization with EPAP valve and group 3 nebulization with NIV bi-level pressure mode. The radioaerosol deposition pattern will be evaluated through Pulmonary Scintigraphy and regional pulmonary ventilation through EIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II (moderate) and III (severe) COPD according to the guidelines of the Global Initiative for Chronic Obstructive Lung Disease (GOLD)

Exclusion Criteria:

* unable to understand or perform procedures that present rheumatic or orthopedic diseases or deformities / abnormalities in the spine that compromise the mechanics of the respiratory system; respiratory comorbidities such as asthma, bronchiectasis and sequela of tuberculosis, cardiovascular and neurological comorbidities; hemodynamic instability defined as heart rate greater than 150 bpm, or systolic pressure less than 90 mmHg; hypertension (blood pressure> 149/89 mmHg) or hypotension (blood pressure <90/60 mmHg) at the time of collection; pregnancy or suspected pregnancy; and any contraindications for the use of PEP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change of Pulmonary Function | 30 minutes after intervention
  Pulmonary function test performed through spirometry
Change of Aerosol deposition in the lungs | Immediately after intervention
  The pulmonary deposition index (PPI), expressed in percentage terms and obtained by the ratio of the number of counts of each ROI to the total number of counts of the respective lung.
Change of Regional pulmonary ventilation | 30 minutes after intervention
  The impedance variation (AZ) and regional pulmonary ventilation (ZEE) will be evaluated for each region of interest.

SECONDARY OUTCOMES:
Change of Ventilatory pattern | 30 minutes after intervention
  Respiratory rate, tidal volume, minute volume, inspiratory time, expiratory time, and total time.
Change of Heart Rate | 30 minutes after intervention
  Heart Rate
Change of Peripheral Oxygen Saturation | Immediately and 30 minutes after intervention
  Peripheral Oxygen Saturation

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Rattes, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Department of Physical Therapy, Federal University of Pernambuco, Recife, Pernambuco, Brazil, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No